CLINICAL TRIAL: NCT04657965
Title: Clinical Trial for the Safety and Efficacy of Sequential of LMP1 CAR-T for Patients With LMP1 Positive Infectious Diseases and Hematological Malignancies
Brief Title: LMP1 CAR-T for Patients With LMP1 Positive Infectious Diseases and Hematological Malignancies
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMP1-001
Record Dates: First submitted 2020-10-22; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Infectious Diseases; Hematological Malignancies
Keywords: Infectious diseases; Hematological Malignancies; CAR T-cell therapy; LMP1
MeSH Terms: conditions — Communicable Diseases; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of LMP1 CAR T-cells (Experimental): Each subject receive LMP1 CAR T-cells by intravenous infusion
  Interventions: Drug: LMP1 CAR T-cells

INTERVENTIONS:
Drug: LMP1 CAR T-cells — Each subject receive LMP1 CAR T-cells by intravenous infusion
  Other Names: LMP1 CAR-T cells injection

SUMMARY:
A study of LMP1 CAR-T for patients with LMP1 positive infectious diseases and hematological malignancies

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for LMP1 positive infectious diseases and hematological malignancies. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 144 patients will be enrolled. Primary objective is to explore the safety, main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

Only applicable to the inclusion criteria of CAEBV

1. Subjects who are diagnosed with CAEBV according to the Okano revised standard proposed by the Japanese Ministry of Health, Labour and Welfare Research Group for the Prevention of Refractory Diseases;
2. All CAEBV patients who have not achieved complete remission, including:

   1. Active phase: EBV-DNA level in PBMC is higher than 1×10^2.5 copies/μg DNA, with symptoms and signs of active diseases such as fever, hepatomegaly, splenomegaly, abnormal liver function, decrease of blood three lines, lymphadenopathy, and progressive skin lesions with increased EBV titer in peripheral blood;
   2. inactive phase: EBV-DNA level in PBMC is higher than 1×10^2.5 copies/μg DNA, without symptoms and signs of active diseases;
3. The disease has not yet progressed to hematopoietic lymphohistiocytosis (HLH);

Only applicable to the inclusion criteria of LMP1-positive ENKTL:

1. According to the 2016 WHO classification criteria for lymphocytic tumors: Subjects diagnosed by histopathology as extranodal NK/T cell lymphoma, nasal type (ENKTL) with LMP1 positive in tumor tissue;
2. R/R ENKTL (meets one of the following prerequisites)

   1. Without remission or with progression after receiving second-line or higher-line chemotherapy/chemotherapy + radiotherapy;
   2. Primary drug resistance;
   3. With recurrence after receiving autologous/allogeneic hematopoietic stem cell transplantation;
3. According to 2014 Lugano standard, there should be at least one evaluable tumor lesion.

Only applicable to the inclusion criteria for LMP1-positive HL:

1. According to the 2016 WHO classification criteria for lymphocytic tumors, subjects with Hodgkin lymphoma diagnosed by histopathology (HD) and LMP1 positive in tumor tissue;
2. R/R HD (meets one of the following prerequisites):

   1. Without remission or with progression after receiving second-line or higher-line chemotherapy;
   2. Primary resistance Drugs;
   3. With recurrence after receiving autologous hematopoietic stem cell transplantation;
3. According to the Lugano 2014 standard, there should be at least one evaluable tumor lesion;

Only applicable to the inclusion criteria for LMP1-positive PTLD:

1. Only PTLD after hematopoietic stem cell transplantation;
2. According to the 2016 WHO classification criteria for lymphocytic tumors, subjects with PTLD diagnosed by histopathology and LMP1 positive in tumor tissue;
3. Excluding PTLD of early-stage
4. R/R PTLD (meets one of the following prerequisites):

   1. Without remission or with progression after receiving rituximab-based standard treatment;
   2. Primary drug resistance;
5. According to the Lugano 2014 standard, there should be at least one evaluable tumor lesion

Exclusion Criteria:

Subjects with any of the following exclusion criteria were not eligible for this trial:

1. History of craniocerebral trauma, conscious disturbance,epilepsy,cerebrovascular ischemia, and cerebrovascular, hemorrhagic diseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
3. Pregnant (or lactating) women;
4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
5. Active infection of hepatitis B virus or hepatitis C virus;
6. Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving in haled steroids;
7. Previously treated with any CAR-T cell product or other genetically modified T cell therapies;
8. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
9. Other uncontrolled diseases that were not suitable for this trial;
10. Patients with HIV infection;
11. Any situations that the investigator believes may increase the risk ofpatients or interfere with the results of study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after LMP1 targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after LMP1 targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Chronic active EB virus infection (CAEBV), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + PR) at Month 1, 3, 6, 12, 18 and 24
CAEBV，Duration of remission（DOR） | Up to 2 years after LMP1 CAR-T cells infusion
  From the first remission after LMP1 CAR-T cells to relapse, death or the last visit
CAEBV, Overall survival (OS) | Up to 2 years after LMP1 CAR-T cells infusion
  From the first infusion of LMP1 CAR-T cells to death or the last visit
CAEBV, Relapse rate(RR) | At Month 6, 12, 18 and 24
  From the first remission after LMP1 CAR-T cells to relapse or the last visit
CAEBV, Event-free survival (EFS) | Up to 2 years after LMP1 CAR-T cells infusion
  From the first infusion of LMP1 CAR-T cells to the occurrence of any event, including death, relapse or gene relapse, disease progression (any one occurs first), and the last visit
Hodgkin's lymphoma(HL), Extranodal NK/T cell lymphoma(ENKTL),Nasal type, Lymphoproliferative disease after hematopoietic stem cell transplantation, (post-HSCT PTLD),Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + PR) at Month 1, 3, 6, 12, 18 and 24
HL, ENKTL, PTLD, OS | Up to 2 years after LMP1 CAR-T cells infusion
  From the first infusion of LMP1 CAR-T cells to death or the last visit
HL, ENKTL, PTLD, EFS | Up to 2 years after LMP3 CAR-T cells infusion
  From the first infusion of LMP1 CAR-T cells to the occurrence of any event, including death, relapse or gene relapse, disease progression (any one occurs first), and the last visit
Quality of life | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale (Barthel Index) [max score: 100, min score: 0, higher scores mean a better outcome] at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale [max score: 56, min score: 14, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Hospital Anxiety and Depression Scale (HADS) [max score: 42, min score: 0, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No